CLINICAL TRIAL: NCT02795429
Title: A Phase Ib/II, Open-label, Multi-center Study of INC280 in Combination With PDR001 or PDR001 Single Agent in Advanced Hepatocellular Carcinoma.
Brief Title: Phase Ib/II Study of INC280 + PDR001 or PDR001 Single Agent in Advanced HCC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC280X2108; 2015-005417-76 (EudraCT Number)
Record Dates: First submitted 2016-05-17; First posted 2016-06-10 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Phase Ib/II; INC280; PDR001; capmatinib; spartalizumab; checkpoint inhibitor; PD-1; Liver cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — spartalizumab; capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W (Experimental): Capmatinib 200 mg administered orally on a continuous twice daily (BID) dosing schedule in combination with spartalizumab 300 mg administered intravenously once every 3 weeks (Q3W) in Phase Ib
  Interventions: Drug: Spartalizumab; Drug: Capmatinib
- Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W (Experimental): Capmatinib 300 mg administered orally on a continuous twice daily (BID) dosing schedule in combination with spartalizumab 300 mg administered intravenously once every 3 weeks (Q3W) in Phase Ib
  Interventions: Drug: Spartalizumab; Drug: Capmatinib
- Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W (Experimental): Capmatinib 400 mg administered orally on a continuous twice daily (BID) dosing schedule in combination with spartalizumab 300 mg administered intravenously once every 3 weeks (Q3W) in Phase Ib
  Interventions: Drug: Spartalizumab; Drug: Capmatinib
- Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W (Experimental): Capmatinib 400 mg administered orally on a continuous twice daily (BID) dosing schedule in combination with spartalizumab 300 mg administered intravenously once every 3 weeks (Q3W) in Phase II
  Interventions: Drug: Spartalizumab; Drug: Capmatinib
- Phase II: Spartalizumab 300 mg Q3W (Experimental): Spartalizumab 300 mg administered intravenously once every 3 weeks (Q3W) in Phase II
  Interventions: Drug: Spartalizumab

INTERVENTIONS:
Drug: Spartalizumab — Spartalizumab administered via intravenous (i.v.) infusion once every 3 weeks (Q3W)
  Other Names: PDR001
Drug: Capmatinib — Capmatinib administered orally as a tablet on a continuous twice daily (BID) dosing schedule
  Other Names: INC280
  Arms: Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W; Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W; Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W; Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W

SUMMARY:
The purpose of this study of capmatinib (INC280) and spartalizumab (PDR001) was to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and antitumor activity of spartalizumab administered intravenously (i.v.) as a single agent or in combination with capmatinib administered orally in adult patients with advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This was a Phase Ib/II, open label, multicenter study starting with a Phase Ib dose escalation part followed by a randomized Phase II part in patients with advanced hepatocellular carcinoma. Capmatinib was administered orally twice daily (BID) and spartalizumab was administered i.v. every 3 weeks (Q3W) until the occurrence of unacceptable toxicity, progressive disease as per irRC and/or treatment was discontinued at the discretion of the Investigator or the participant. A complete cycle of treatment was defined as 21 days.

During the Phase Ib dose escalation part of the study, participants were treated with capmatinib in combination with a fixed dose of spartalizumab until the maximum tolerated dose (MTD) was reached or the recommended phase 2 dose (RP2D) was established. The capmatinib dose was increased and the spartalizumab dose remained constant.

Once the MTD and/or RP2D were declared for capmatinib in combination with spartalizumab, additional participants were enrolled in the Phase II part in order to assess the anti-tumor activity of capmatinib in combination with spartalizumab and spartalizumab single agent. Participants were randomly assigned, in a 1:1 ratio, to treatment with either capmatinib in combination with spartalizumab or spartalizumab single agent.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented locally advanced recurrent or metastatic HCC or for patients with cirrhosis according to the American Association for the Study of Liver Diseases (AASLD) and Asian Pacific Association for the study of the liver (APASL) criteria. Current cirrhotic status of Child Pugh Class A (5-6 points), with no encephalopathy and/or clinically significant ascites (defined as requiring the use of diuretics or paracentesis treatment).
2. Patients must have received prior systemic sorafenib treatment for HCC with documented progression during or after discontinuation of sorafenib treatment (for France only: patients must have received at least 8 weeks of prior sorafenib treatment), or are intolerant to sorafenib (defined as documented Grade 3 or 4 adverse events that led to sorafenib discontinuation),.
3. ECOG Performance Status ≤ 1.
4. Willing and able to swallow and retain oral medication.

Exclusion Criteria:

1. Use of any live vaccines within 4 weeks of initiation of study treatment.
2. History of severe hypersensitivity reactions to other monoclonal antibodies (mAbs).
3. Clinically significant pleural effusion that either required pleurocentesis or is associated with shortness of breath.
4. Active autoimmune disease or a documented history of autoimmune disease.
5. Clinically significant, uncontrolled heart diseases.
6. Patient having out of range laboratory values defined as:

   * Total bilirubin > 2 mg/dL, except for patients with Gilbert's syndrome who are excluded if total bilirubin > 3.0 x ULN or direct bilirubin > 1.5 x ULN
   * Alanine aminotransferase (ALT) > 5 x ULN
   * Aspartate aminotransferase (AST) > 5 x ULN
   * Coagulation: Prothrombin Time (PT) > 4 seconds more than the ULN or International Normalized Ratio (INR) > 1.7
   * Absolute neutrophil count (ANC) < 1.5 x 109/L
   * Platelet count < 75 x 109/L
   * Hemoglobin < 9 g/dL
   * Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) < 45 mL/min
   * Asymptomatic serum amylase grade > 2 (1.5-2.0 x ULN). Patients with grade 1 or grade 2 serum amylase at the beginning of the study must be confirmed to have no signs or symptoms suggesting pancreatitis or pancreatic injury (e.g., elevated P-amylase, abnormal imaging findings of pancreas, etc.)
   * Serum lipase > ULN
   * Potassium, Magnesium, Phosphorus, total Calcium (corrected for serum albumin) outside of normal limits (patients may be enrolled if corrected to within normal limits with supplements during screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- China (2):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
- France (3):
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
- Novartis Investigative Site, Seoul, South Korea
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Santoro A, Assenat E, Yau T, Delord JP, Maur M, Knox J, Cattan S, Lee KH, Del Conte G, Springfeld C, Leo E, Xyrafas A, Fairchild L, Mardjuadi F, Chan SL. A phase Ib/II trial of capmatinib plus spartalizumab vs. spartalizumab alone in patients with pretreated hepatocellular carcinoma. JHEP Rep. 2024 Jan 28;6(4):101021. doi: 10.1016/j.jhepr.2024.101021. eCollection 2024 Apr. PMID 38617599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 18 investigative sites in 8 countries.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. Screening evaluations were performed within 21 days prior to the first dose of study medication. After screening, the treatment period started on Cycle 1 Day 1.
Period: Overall Study
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Started | 6 | 10 | 11 | 32 | 30
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 10 | 11 | 32 | 30
Not completed — Adverse Event | 1 | 2 | 1 | 2 | 1
Not completed — Death | 1 | 0 | 1 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 2 | 1 | 5
Not completed — Progressive disease | 3 | 7 | 6 | 26 | 20
Not completed — Subject/guardian decision | 1 | 1 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W | Total
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (7.42) | 63.2 (10.24) | 64.6 (8.99) | 64.8 (10.02) | 63.4 (9.97) | 64.4 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 3 | 5 | 12
  Male | 6 | 8 | 9 | 29 | 25 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 3 | 4 | 12 | 12 | 34
  White | 3 | 7 | 6 | 10 | 10 | 36
  Unknown | 0 | 0 | 1 | 10 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-treatment Period
Description: Number of participants with AEs and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
  AE grades to characterize the severity of the AEs were based on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. For CTCAE v4.03, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE.
  The on-treatment period is defined from the day of first administration of study treatment up to 30 days after the date of its last administration.
Time Frame: From first dose of study medication up to 30 days after last dose, with a maximum duration of 3.3 years
Population: All patients who had received at least one dose of spartalizumab or capmatinib in the Phase Ib part
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11
Participants
  AEs | 6 | 10 | 10
  Treatment-related AEs | 5 | 7 | 10
  AEs with grade ≥ 3 | 6 | 7 | 7
  Treatment-related AEs with grade ≥ 3 | 4 | 4 | 6
  SAEs | 1 | 1 | 6
  Treatment-related SAEs | 0 | 0 | 5
  Fatal SAEs | 1 | 0 | 1
  Treatment-related fatal SAEs | 0 | 0 | 1
  AEs leading to discontinuation | 3 | 4 | 4
  Treatment-related AEs leading to discontinuation | 2 | 1 | 4
  AEs leading to dose adjustment/interruption | 3 | 6 | 7
  AEs requiring additional therapy | 6 | 9 | 10
  AE due to infusion reaction | 0 | 0 | 1

2. Primary Outcome: Phase Ib: Number of Participants With Dose-Limiting Toxicities (DLTs) During the First 2 Cycles of Treatment
Description: A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, inter-current illness or concomitant medications that occurs within the first 2 cycles of treatment with capmatinib in combination with spartalizumab during the dose escalation part of the study. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher. The duration of one treatment cycle is 21 days.
Time Frame: 42 days
Population: Patients in Phase Ib who either met the minimum exposure criterion and had sufficient safety evaluations, or had experienced a DLT during Cycles 1 and 2. A patient was considered to have met the minimum exposure criterion if received at least 2 doses of spartalizumab and 28 days of capmatinib during Cycles 1 and 2. Patients who did not experience a DLT during the first 2 cycles were considered to have sufficient safety evaluations if they had been observed for at least 42 days after first dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 8 | 9
Participants | 0 | 0 | 1

3. Primary Outcome: Phase Ib: Number of Participants With Dose Reductions and Dose Interruptions of Capmatinib and Spartalizumab
Description: Number of participants with at least one dose reduction of capmatinib and spartalizumab and number of participants with at least one dose interruption of capmatinib and spartalizumab.
  No dose modifications (i.e. dose reduction) were allowed for spartalizumab.
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 3.2 years
Population: All patients who had received at least one dose of spartalizumab or capmatinib in the Phase Ib part
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11
Participants
  Capmatinib dose reduction | 2 | 4 | 8
  Capmatinib dose interruption | 4 | 6 | 8
  Spartalizumab dose reduction | 0 | 0 | 0
  Spartalizumab dose interruption | 4 | 4 | 7

4. Primary Outcome: Phase Ib: Dose Intensity of Capmatinib
Description: Dose intensity of capmatinib was calculated as actual cumulative dose in milligrams divided by duration of exposure in days.
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 3.2 years
Population: All patients who had received at least one dose of spartalizumab or capmatinib in the Phase Ib part
Measure: Median (Full Range); unit: mg/day
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11
mg/day | 391.2 [294 to 400] | 580.0 [390 to 600] | 755.6 [371 to 800]

5. Primary Outcome: Phase Ib: Dose Intensity of Spartalizumab
Description: Dose intensity of spartalizumab was calculated as actual cumulative dose in milligrams divided by duration of exposure in weeks and then multiplied by 3 weeks (3W).
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 3.2 years
Population: All patients who had received at least one dose of spartalizumab or capmatinib in the Phase Ib part
Measure: Median (Full Range); unit: mg/3W
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11
mg/3W | 293.18 [235.7 to 300.0] | 300.00 [225.0 to 300.0] | 300.00 [272.7 to 300.0]

6. Primary Outcome: Phase II: Overall Response Rate (ORR) Per RECIST v1.1
Description: Tumor response was based on local investigator assessment as per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. ORR per RECIST v1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From start of treatment until end of treatment, assessed up to 2.2 years
Population: All patients to whom study treatment was assigned by randomization in the Phase II part
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 32 | 30
percentage of participants | 9.4 [2.0 to 25.0] | 10.0 [2.1 to 26.5]
Statistical Analysis 1: Comparison: Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W vs Phase II: Spartalizumab 300 mg Q3W; Test type: Superiority; Bayesian Logistic Regression Model; Odds Ratio (OR) = 0.561 — Posterior probability that the odds ratio (ORRspartalizumab +capmatinib to ORRspartalizumab) was ≥ 1

7. Secondary Outcome: Phase Ib and Phase II: Best Overall Response (BOR) Per RECIST v1.1
Description: BOR is defined as the best response recorded from the start of the study treatment until disease progression/recurrence, based on local investigator assessment per RECIST v1.1.
  For RECIST v1.1, R=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters; PD= At least a 20% increase in the sum of diameters of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition, the sum must also demonstrate an absolute increase of at least 5 mm; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression).
  The number of participants in each response category is reported in the table.
Time Frame: From start of treatment until end of treatment, assessed up to 3.2 years in Phase Ib and up to 2.2 years in Phase II
Population: All patients who received at least one dose of study treatment in the Phase Ib part, and all patients to whom study treatment was assigned by randomization in the Phase II part.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 2 | 0 | 2 | 3 | 3
  Stable Disease (SD) | 1 | 7 | 2 | 12 | 9
  Progressive Disease (PD) | 3 | 2 | 7 | 13 | 15
  Unknown | 0 | 1 | 0 | 4 | 3

8. Secondary Outcome: Phase Ib and Phase II: Best Overall Response (BOR) Per irRC
Description: BOR is defined as the best response recorded from the start of the study treatment until disease progression/recurrence, based on local investigator assessment per Immune-related Response Criteria (irRC).
  For irRC, irCR=Disappearance of all non-nodal target lesions and non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; irPR= At least a 30% decrease in the sum of diameters of all target lesions including new measurable lesions, taking as reference the baseline sum of diameters; irPD= At least a 20% increase in the sum of diameters of all measured target lesions including new measurable lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition, the sum must also demonstrate an absolute increase of at least 5 mm; irSD= Neither sufficient shrinkage to qualify for irPR or irCR nor an increase in lesions which would qualify for irPD).
Time Frame: From start of treatment until end of treatment, assessed up to 3.2 years in Phase Ib and up to 2.2 years in Phase II
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
Participants
  Immune-related Complete Response (irCR) | 0 | 0 | 0 | 0 | 0
  Immune-related Partial Response (irPR) | 2 | 0 | 3 | 4 | 3
  Immune-related Stable Disease (irSD) | 1 | 7 | 3 | 15 | 9
  Immune-related Progressive Disease (irPD) | 3 | 2 | 5 | 10 | 14
  Unknown | 0 | 1 | 0 | 3 | 4

9. Secondary Outcome: Phase Ib: Overall Response Rate (ORR) Per RECIST v1.1
Description: Tumor response was based on local investigator assessment as per RECIST v1.1. ORR per RECIST v1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From start of treatment until end of treatment, assessed up to 3.2 years
Population: All patients who had received at least one dose of spartalizumab or capmatinib capmatinib in the Phase Ib part
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11
percentage of participants | 33.3 [4.3 to 77.7] | 0 [0.0 to 30.8] | 18.2 [2.3 to 51.8]

10. Secondary Outcome: Phase Ib and Phase II: Overall Response Rate (ORR) Per irRC
Description: Tumor response was based on local investigator assessment as per irRC. ORR per irRC is defined as the percentage of participants with a best overall response of immune related Complete Response (irCR) or immune related Partial Response (irPR).
  For irRC, irCR=Disappearance of all non-nodal target lesions and non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; irPR= At least a 30% decrease in the sum of diameters of all target lesions including new measurable lesions, taking as reference the baseline sum of diameters.
Time Frame: From start of treatment until end of treatment, assessed up to 3.2 years in Phase Ib and up to 2.2 years in Phase II
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
percentage of participants | 33.3 [4.3 to 77.7] | 0 [0.0 to 30.8] | 27.3 [6.0 to 61.0] | 12.5 [3.5 to 29.0] | 10.0 [2.1 to 26.5]

11. Secondary Outcome: Phase Ib and Phase II: Duration of Response (DOR) Per RECIST v1.1
Description: DOR only applies to patients for whom best overall response is complete response (CR) or partial response (PR) based on local investigator assessment of overall lesion response according to RECIST v1.1. DOR is defined as the time from the date of first documented response (confirmed CR or confirmed PR) to the date of first documented disease progression or death due to any cause. If a patient not had an event, duration was censored at the date of last adequate tumor assessment before the start of a new anticancer therapy, if any.
  According to the statistical analysis plan (SAP), summary estimates of DOR using the Kaplan-Meier method were planned to be reported if there were at least 10 patients achieving a confirmed CR or PR in each treatment group/arm.
Time Frame: From first documented response to first documented disease progression or death due to any cause, assessed up to 3.2 years in Phase Ib and up to 2.2 years in Phase II
Population: All participants in Phase Ib and II for whom best overall response is complete response (CR) or partial response (PR) as per RECIST v1.1 based on local investigator assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 2 | 0 | 2 | 3 | 3
months | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. |  | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP.

12. Secondary Outcome: Phase Ib and Phase II: Duration of Response (DOR) Per irRC
Description: DOR only applies to patients for whom best overall response is immune-related complete response (irCR) or immune-related partial response (irPR) based on local investigator assessment of overall lesion response according to irRC. DOR is defined as the time from the date of first documented response (confirmed irCR or confirmed irPR) to the date of first documented disease progression or death due to any cause. If a patient not had an event, duration was censored at the date of last adequate tumor assessment before the start of a new anticancer therapy, if any.
  According to the statistical analysis plan (SAP), summary estimates of DOR using the Kaplan-Meier method were planned to be reported if there were at least 10 patients achieving a confirmed irCR or irPR in each treatment group/arm.
Time Frame: as for outcome 11
Population: All participants in Phase Ib and II for whom best overall response is immune-related complete response (irCR) or immune-related partial response (irPR) as per irRC based on local investigator assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 2 | 0 | 3 | 4 | 3
months | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. |  | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP.

13. Secondary Outcome: Phase Ib and Phase II: Time to Response (TTR) Per RECIST v1.1
Description: TTR is defined as the time from the date of start of treatment to the date of first documented response (CR or PR, which must be confirmed subsequently) for patients who achieved a confirmed CR or PR. Tumor response was based on local investigator assessment per RECIST v1.1.
  Patients who did not achieve a confirmed CR or PR were censored at the maximum follow-up time for patients who had a Progression-Free Survival (PFS) event (i.e. either progressed or died due to any cause), or at the date of last adequate tumor assessment before the start of a new anticancer therapy (if any) otherwise.
  According to the statistical analysis plan (SAP), summary estimates of TTR using the Kaplan-Meier method were planned to be reported if there were at least 10 patients achieving a confirmed CR or PR in each treatment group/arm.
Time Frame: From start of treatment until first documented response, assessed up to 3.2 years in Phase Ib and up to 2.2 years in Phase II
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
months | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP.

14. Secondary Outcome: Phase Ib and Phase II: Time to Response (TTR) Per irRC
Description: TTR is defined as the time from the date of start of treatment to the date of first documented response (irCR or irPR, which must be confirmed subsequently) for patients who achieved a confirmed irCR or irPR. Tumor response was based on local investigator assessment per irRC.
  Patients who did not achieve a confirmed irCR or irPR were censored at the maximum follow-up time for patients who had a Progression-Free Survival (PFS) event (i.e. either progressed or died due to any cause), or at the date of last adequate tumor assessment before the start of a new anticancer therapy (if any) otherwise.
  According to the statistical analysis plan (SAP), summary estimates of TTR using the Kaplan-Meier method were planned to be reported if there were at least 10 patients achieving a confirmed irCR or irPR in each treatment group/arm.
Time Frame: as for outcome 13
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
months | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP.

15. Secondary Outcome: Phase Ib and Phase II: Progression-Free Survival (PFS) Per RECIST v1.1
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression per RECIST v1.1 or death due to any cause. If a patient did not experience an event or started a new anticancer therapy, PFS was censored at the date of the last adequate tumor evaluation before the start of a new anticancer therapy, if any. Tumor response was based on local investigator assessment per RECIST v1.1.
  PFS was estimated using the Kaplan-Meier Method.
Time Frame: From start of treatment until first documented progression or death due to any cause, assessed up to 3.2 years in Phase Ib and up to 2.2 years in Phase II
Population: All patients who received at least one dose of study treatment in the Phase Ib part, and all patientss to whom study treatment was assigned by randomization in the Phase II part.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
months | 3.42 [1.18 to NA] — Not estimable due to insufficient number of participants with events. | 4.44 [1.25 to NA] — Not estimable due to insufficient number of participants with events. | 1.35 [1.22 to 13.73] | 2.79 [2.60 to 3.88] | 2.79 [1.45 to 4.07]

16. Secondary Outcome: Phase Ib and Phase II: Progression-Free Survival (PFS) Per irRC
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented and confirmed progression per irRC or death due to any cause. If a patient did not experience an event or started a new anticancer therapy, PFS was censored at the date of the last adequate tumor evaluation before the start of a new anticancer therapy, if any. Tumor response was based on local investigator assessment per irRC.
  PFS was estimated using the Kaplan-Meier Method.
Time Frame: as for outcome 15
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
months | 3.42 [1.18 to NA] — Not estimable due to insufficient number of participants with events. | 4.44 [1.68 to NA] — Not estimable due to insufficient number of participants with events. | 5.55 [1.25 to NA] — Not estimable due to insufficient number of participants with events. | 3.06 [2.63 to 4.17] | 2.79 [1.61 to 5.75]

17. Secondary Outcome: Phase Ib and Phase II: Time to Progression (TTP) Per RECIST v1.1
Description: TTP is defined as the time from the date of start of treatment to the date of the first documented progression per RECIST v1.1 or death due to underlying cancer. If a patient did not experience an event or started a new anticancer therapy, TTP was censored at the date of the last adequate tumor evaluation before the start of a new anticancer therapy, if any. Tumor response was based on local investigator assessment per RECIST v1.1.
  TTP was estimated using the Kaplan-Meier Method.
Time Frame: From start of treatment until first documented progression or death due to underlying cancer, assessed up to 3.2 years in Phase Ib and up to 2.2 years in Phase II
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
months | 3.42 [1.18 to NA] — Not estimable due to insufficient number of participants with events. | 4.44 [1.25 to NA] — Not estimable due to insufficient number of participants with events. | 1.35 [1.22 to NA] — Not estimable due to insufficient number of participants with events. | 2.79 [2.60 to 3.88] | 2.79 [1.45 to 4.07]

18. Secondary Outcome: Phase Ib and Phase II: Time to Progression (TTP) Per irRC
Description: TTP is defined as the time from the date of start of treatment to the date of the first documented and confirmed progression per irRC or death due to underlying cancer. If a patient did not experience an event or started a new anticancer therapy, TTP was censored at the date of the last adequate tumor evaluation before the start of a new anticancer therapy, if any. Tumor response was based on local investigator assessment per irRC.
Time Frame: as for outcome 17
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
months | 3.42 [1.18 to NA] — Not estimable due to insufficient number of participants with events. | 4.44 [1.68 to NA] — Not estimable due to insufficient number of participants with events. | 5.55 [1.25 to NA] — Not estimable due to insufficient number of participants with events. | 3.06 [2.63 to 4.17] | 2.79 [1.61 to 5.75]

19. Secondary Outcome: Phase Ib and Phase II: Overall Survival (OS)
Description: OS is defined as the time from date of start of treatment to date of death due to any cause. If a patient was not known to have died, OS time was censored at the date of last contact.
  OS was estimated using the Kaplan-Meier Method.
Time Frame: From start of treatment until death due to any cause, assessed up to 3.6 years in Phase Ib and up to 2.9 years in Phase II
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
months | 14.98 [2.37 to NA] — Not estimable due to insufficient number of participants with events. | 12.11 [1.68 to 19.45] | 16.53 [2.83 to NA] — Not estimable due to insufficient number of participants with events. | 14.88 [9.00 to 19.48] | 9.78 [3.65 to 22.31]

20. Secondary Outcome: Phase II: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-treatment Period
Description: as for outcome 1
Time Frame: From first dose of study medication up to 30 days after last dose, with a maximum duration of 2.3 years
Population: All patients to whom study treatment was assigned by randomization in the Phase II part
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 32 | 30
Participants
  AEs | 32 | 30
  Treatment-related AEs | 30 | 18
  AEs with grade ≥ 3 | 25 | 15
  Treatment-related AEs with grade ≥ 3 | 18 | 3
  SAEs | 14 | 10
  Treatment-related SAEs | 7 | 1
  Fatal SAEs | 1 | 1
  AEs leading to discontinuation | 10 | 1
  Treatment-related AEs leading to discontinuation | 7 | 0
  AEs leading to dose adjustment/interruption | 22 | 11
  AEs requiring additional therapy | 30 | 29
  AE due to infusion reaction | 1 | 0

21. Secondary Outcome: Phase II: Number of Participants With Dose Reductions and Dose Interruptions of Capmatinib and Spartalizumab
Description: as for outcome 3
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 2.2 years
Population: All patients to whom study treatment was assigned by randomization in the Phase II part
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 32 | 30
Participants
  Capmatinib dose reduction: number analyzed (Participants) | 32 | 0
  Capmatinib dose reduction | 18 |
  Capmatinib dose interruption: number analyzed (Participants) | 32 | 0
  Capmatinib dose interruption | 22 |
  Spartalizumab dose reduction | 0 | 0
  Spartalizumab dose interruption | 12 | 13

22. Secondary Outcome: Phase II: Dose Intensity of Capmatinib
Description: as for outcome 4
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 2.2 years
Population: All patients assigned by randomization to capmatinib in combination with spartalizumab in the Phase II part
Measure: Median (Full Range); unit: mg/day
Arm/Group | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 32 | 0
mg/day | 696.4 [167 to 800] |

23. Secondary Outcome: Phase II: Dose Intensity of Spartalizumab
Description: as for outcome 5
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 2.2 years
Population: All patients to whom study treatment was assigned by randomization in the Phase II part
Measure: Median (Full Range); unit: mg/3W
Arm/Group | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 32 | 30
mg/3W | 300.00 [200.0 to 300.0] | 300.00 [166.7 to 300.0]

24. Secondary Outcome: Phase Ib: Maximum Observed Plasma Concentration (Cmax) of Capmatinib
Description: Pharmacokinetic (PK) parameters were calculated based on capmatinib plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed plasma concentration following a dose.
Time Frame: pre-dose, 0.5, 1, 2, 4 and 8 hours post capmatinib dose on Cycle 2 Day 1 (C2D1). The duration of one cycle was 21 days.
Population: All patients in Phase Ib who provided an evaluable capmatinib PK profile on C2D1. Capmatinib PK profile was considered evaluable if all the following conditions were satisfied: patient took the same dose of capmatinib for at least 3 consecutive days prior to sampling, patient had the pre-dose sample collected before next dose administration and at least 9 hours after last dose administration, patient did not vomit within 4 hours after dosing and patient provided at least 1 primary PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 4 | 5 | 7
ng/mL | 1680 (64.0) | 3110 (61.2) | 4980 (23.0)

25. Secondary Outcome: Phase Ib: Time to Reach Maximum Plasma Concentration (Tmax) of Capmatinib
Description: Pharmacokinetic (PK) parameters were calculated based on capmatinib plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) plasma concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: pre-dose, 0.5, 1, 2, 4 and 8 hours post capmatinib dose on Cycle 2 Day 1 (C2D1). The duration of one cycle was 21 days.
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 4 | 5 | 7
hours | 0.959 [0.567 to 1.00] | 1.00 [1.00 to 2.05] | 1.00 [1.00 to 4.22]

26. Secondary Outcome: Phase Ib: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Capmatinib
Description: Pharmacokinetic (PK) parameters were calculated based on capmatinib plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: pre-dose, 0.5, 1, 2, 4 and 8 hours post capmatinib dose on Cycle 2 Day 1 (C2D1). The duration of one cycle was 21 days.
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 4 | 5 | 7
hours*ng/mL | 5740 (51.6) | 8570 (60.7) | 16000 (30.6)

27. Secondary Outcome: Phase II: Pre-dose Plasma Concentration of Capmatinib
Description: Capmatinib plasma concentration was assessed in samples taken at pre-dose. Pre-dose samples were collected before the next dose administration.
Time Frame: Pre-dose of capmatinib on Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 and Cycle 6 Day 1. The duration of one cycle was 21 days.
Population: All patients in Phase II part who provided an evaluable capmatinib concentration at the specified timepoints. Capmatinib concentration was considered evaluable if all the following conditions were satisfied: patient took the same dose of capmatinib for at least 3 consecutive days prior to sampling, patient had the pre-dose sample collected before next dose administration and at least 9 hours after last dose administration, patient did not vomit within 4 hours after the dosing prior to sampling.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 32 | 0
ng/mL
  Cycle 2 Day 1: number analyzed (Participants) | 16 | 0
  Cycle 2 Day 1 | 607 (99.4) |
  Cycle 3 Day 1: number analyzed (Participants) | 16 | 0
  Cycle 3 Day 1 | 345 (110) |
  Cycle 4 Day 1: number analyzed (Participants) | 16 | 0
  Cycle 4 Day 1 | 410 (132) |
  Cycle 5 Day 1: number analyzed (Participants) | 10 | 0
  Cycle 5 Day 1 | 363 (68.6) |
  Cycle 6 Day 1: number analyzed (Participants) | 11 | 0
  Cycle 6 Day 1 | 275 (102) |

28. Secondary Outcome: Phase Ib and Phase II: Maximum Observed Serum Concentration (Cmax) of Spartalizumab
Description: Pharmacokinetic (PK) parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
Time Frame: pre-dose, 1, 24, 48, 72, 168, 240, 336 and 504 hours after completion of spartalizumab infusion on Cycle 1 and Cycle 3. The duration of one cycle was 21 days.
Population: All patients in Phase Ib and Phase II who provided an evaluable PK profile of spartalizumab on Cycle 1 and Cycle 3. The spartalizumab PK profile was considered evaluable if all the following conditions were satisfied: patient received the planned treatment with spartalizumab and patient provided at least 1 primary PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
µg/mL
  Cycle 1: number analyzed (Participants) | 6 | 9 | 11 | 32 | 30
  Cycle 1 | 75.7 (22.6) | 77.2 (20.9) | 84.7 (23.3) | 81.7 (30.1) | 72.8 (30.9)
  Cycle 3: number analyzed (Participants) | 5 | 8 | 7 | 27 | 21
  Cycle 3 | 105 (35.8) | 101 (22.3) | 128 (20.9) | 115 (30.2) | 101 (42.2)

29. Secondary Outcome: Phase Ib and Phase II: Time to Reach Maximum Serum Concentration (Tmax) of Spartalizumab
Description: Pharmacokinetic (PK) parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 28
Population: All patients in Phase Ib and Phase II who provided an evaluable PK profile of spartalizumab on Cycle 1 Day 1 and Cycle 3 Day 1. The spartalizumab PK profile was considered evaluable if all the following conditions were satisfied: patient received the planned treatment with spartalizumab and patient provided at least 1 primary PK parameter.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
hours
  Cycle 1: number analyzed (Participants) | 6 | 9 | 11 | 32 | 30
  Cycle 1 | 1.51 [1.42 to 1.77] | 1.50 [0.583 to 1.67] | 1.50 [1.18 to 1.73] | 1.64 [0.917 to 581] | 1.59 [0.633 to 22.9]
  Cycle 3: number analyzed (Participants) | 5 | 8 | 7 | 27 | 21
  Cycle 3 | 1.53 [1.50 to 1.60] | 1.47 [1.42 to 22.6] | 1.52 [1.45 to 1.92] | 1.75 [0.00 to 24.2] | 1.58 [1.33 to 22.3]

30. Secondary Outcome: Phase Ib and Phase II: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Spartalizumab
Description: Pharmacokinetic (PK) parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: as for outcome 28
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/mL
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
day*µg/mL
  Cycle 1: number analyzed (Participants) | 6 | 9 | 11 | 32 | 30
  Cycle 1 | 739 (24.7) | 726 (20.9) | 813 (19.4) | 805 (33.4) | 693 (35.3)
  Cycle 3: number analyzed (Participants) | 5 | 8 | 7 | 27 | 21
  Cycle 3 | 1280 (39.2) | 1220 (25.5) | 1630 (23.2) | 1330 (41.6) | 883 (79.1)

31. Secondary Outcome: Phase Ib and Phase II: Percent Marker Area for CD8 Expression in Tumor Samples
Description: The expression of CD8 was measured in tumor samples by immunohistochemical methods. This record summarizes the percent marker area for CD8 expression in tumor samples.
Time Frame: Baseline (screening) and post-baseline (assessed throughout the treatment up to maximum 115 days).
Population: All patients who received at least one dose of study treatment in the Phase Ib part and had a valid assessment for the outcome measure, and all patients to whom study treatment was assigned by randomization in the Phase II part and had a valid assessment for the outcome measure.
Measure: Median (Full Range); unit: CD8 percent marker area
Units Other Than Participants: Tumor samples
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 4 | 9 | 8 | 22 | 23
Number analyzed (Tumor samples) | 5 | 15 | 10 | 29 | 31
CD8 percent marker area
  Baseline: number analyzed (Participants) | 4 | 7 | 7 | 19 | 19
  Baseline: number analyzed (Tumor samples) | 4 | 7 | 7 | 19 | 19
  Baseline | 0.6 [0 to 1] | 0.9 [0 to 37] | 0.4 [0 to 3] | 0.5 [0 to 5] | 0.3 [0 to 27]
  Post-baseline: number analyzed (Participants) | 1 | 8 | 3 | 10 | 12
  Post-baseline: number analyzed (Tumor samples) | 1 | 8 | 3 | 10 | 12
  Post-baseline | 3.0 [3 to 3] | 2.6 [0 to 14] | 1.0 [0 to 1] | 1.3 [0 to 7] | 0.9 [0 to 21]

32. Secondary Outcome: Phase Ib and Phase II: PD-L1 Percent Positive Tumor
Description: The expression of programmed cell death-ligand 1 (PD-L1) was measured in tumor samples by immunohistochemical methods. This record summarizes the PD-L1 positivity percentage in tumor samples.
Time Frame: Baseline (screening) and post-baseline (assessed throughout the treatment up to maximum 115 days).
Population: as for outcome 31
Measure: Median (Full Range); unit: PD-L1 positivity percentage
Units Other Than Participants: Tumor samples
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 4 | 10 | 8 | 26 | 24
Number analyzed (Tumor samples) | 6 | 16 | 10 | 31 | 32
PD-L1 positivity percentage
  Baseline: number analyzed (Participants) | 4 | 8 | 7 | 21 | 22
  Baseline: number analyzed (Tumor samples) | 4 | 8 | 7 | 21 | 22
  Baseline | 0.0 [0 to 5] | 0.0 [0 to 90] | 0.0 [0 to 2] | 0.0 [0 to 7] | 0.0 [0 to 3]
  Post-baseline: number analyzed (Participants) | 2 | 8 | 3 | 10 | 10
  Post-baseline: number analyzed (Tumor samples) | 2 | 8 | 3 | 10 | 10
  Post-baseline | 12.5 [0 to 25] | 0.0 [0 to 100] | 0.0 [0 to 5] | 0.0 [0 to 3] | 0.0 [0 to 5]

33. Post Hoc Outcome: Phase Ib and Phase II: All-Collected Deaths
Description: On-treatment and post-treatment safety follow-up deaths were collected from first dose of study medication to 150 days after the last dose of study medication.
  Post-treatment survival follow-up deaths were collected from day 151 after last dose of study medication to end of study.
  All deaths refer to the sum of on-treatment and post-treatment safety follow-up deaths plus post-treatment survival follow-up deaths.
Time Frame: On-treatment and post-treatment safety follow-up deaths: up to 3.6 years in Phase Ib and 2.6 years in Phase II. Post treatment survival follow-up deaths: up to 3.6 years in Phase Ib and 2.9 years in Phase II.
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W | Phase II: Spartalizumab 300 mg Q3W
Number analyzed (Participants) | 6 | 10 | 11 | 32 | 30
participants
  On-treatment and post-treatment safety follow-up deaths | 3 | 3 | 4 | 8 | 13
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 3 | 7 | 7 | 24 | 17
  Post-treatment survival follow-up deaths | 3 | 5 | 4 | 15 | 10
  All deaths | 6 | 8 | 8 | 23 | 23

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment to 150 days after last dose of study medication (on-treatment and post-treatment safety follow-up), up to 3.6 years in Phase Ib and 2.6 years in Phase II. Deaths were collected in the post treatment survival follow up from 151 days after last dose of study medication until the end of the study, up to 3.6 years in Phase Ib and 2.9 years in Phase II. These are not considered AEs
Description: Any sign or symptom that occurs during the on-treatment and safety follow-up periods. Deaths in the post treatment survival follow-up are not considered Adverse Events.
Groups:
- Phase Ib: Capmatinib 200mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU: AEs during on-treatment period and post-treatment safety follow-up (FU) (up to 150 days post-treatment)
- Phase Ib: Capmatinib 300mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU; Phase Ib: Capmatinib 400mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU; Phase II: Capmatinib 400mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU; Phase II: Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU: AEs during on-treatment period and post-treatment safety follow-up (up to 150 days post-treatment)
- Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU; Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU; Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU; Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU; Phase II: Spartalizumab 300 mg Q3W - Post-treatment Survival FU: Deaths collected in the post-treatment survival follow-up period (starting from day 151 post- treatment). No AEs were collected during this period
Arm/Group | Phase Ib: Capmatinib 200mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU | Phase Ib: Capmatinib 300mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU | Phase Ib: Capmatinib 400mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU | Phase II: Capmatinib 400mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU | Phase II: Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU | Phase II: Spartalizumab 300 mg Q3W - Post-treatment Survival FU
All-Cause Mortality (participants affected / at risk) | 3/6 | 3/10 | 4/11 | 8/32 | 13/30 | 3/3 | 5/7 | 4/7 | 15/24 | 10/17
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/10 | 6/11 | 14/32 | 12/30 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 10/10 | 10/11 | 32/32 | 30/30 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib: Capmatinib 200mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU (N=6) | Phase Ib: Capmatinib 300mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU (N=10) | Phase Ib: Capmatinib 400mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU (N=11) | Phase II: Capmatinib 400mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU (N=32) | Phase II: Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU (N=30) | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU (N=0) | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU (N=0) | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU (N=0) | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU (N=0) | Phase II: Spartalizumab 300 mg Q3W - Post-treatment Survival FU (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 1 | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Haemoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 1 | 0 | 0 | 3 | 2 | NA | NA | NA | NA | NA
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | NA | NA | NA | NA | NA
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Blood corticotrophin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib: Capmatinib 200mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU (N=6) | Phase Ib: Capmatinib 300mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU (N=10) | Phase Ib: Capmatinib 400mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU (N=11) | Phase II: Capmatinib 400mg BID + Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU (N=32) | Phase II: Spartalizumab 300mg Q3W - On-treatment and Post-treatment Safety FU (N=30) | Phase Ib: Capmatinib 200 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU (N=0) | Phase Ib: Capmatinib 300 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU (N=0) | Phase Ib: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU (N=0) | Phase II: Capmatinib 400 mg BID + Spartalizumab 300 mg Q3W - Post-treatment Survival FU (N=0) | Phase II: Spartalizumab 300 mg Q3W - Post-treatment Survival FU (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 4 | 3 | NA | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 3 | 1 | NA | NA | NA | NA | NA
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 1 | 1 | NA | NA | NA | NA | NA
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 1 | 3 | NA | NA | NA | NA | NA
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Diplopia (Eye disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2 | 4 | 3 | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 3 | 7 | 5 | NA | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 2 | 5 | 3 | NA | NA | NA | NA | NA
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Aptyalism (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 1 | 2 | 0 | 7 | 5 | NA | NA | NA | NA | NA
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 3 | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3 | 10 | 6 | NA | NA | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 4 | NA | NA | NA | NA | NA
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | NA | NA | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 2 | 2 | 5 | 15 | 2 | NA | NA | NA | NA | NA
Plicated tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 1 | 4 | 0 | 2 | 2 | NA | NA | NA | NA | NA
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3 | 9 | 1 | NA | NA | NA | NA | NA
Asthenia (General disorders) | 2 | 0 | 2 | 14 | 10 | NA | NA | NA | NA | NA
Chills (General disorders) | 0 | 0 | 2 | 5 | 0 | NA | NA | NA | NA | NA
Fatigue (General disorders) | 2 | 3 | 4 | 4 | 2 | NA | NA | NA | NA | NA
Influenza like illness (General disorders) | 1 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Malaise (General disorders) | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Nodule (General disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 2 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 4 | 6 | 6 | 15 | 6 | NA | NA | NA | NA | NA
Pain (General disorders) | 0 | 1 | 0 | 1 | 2 | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 3 | 0 | 4 | 14 | 5 | NA | NA | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Abscess neck (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | NA | NA | NA | NA | NA
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | NA | NA | NA | NA | NA
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | NA | NA | NA | NA | NA
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | NA | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | NA | NA | NA | NA | NA
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 3 | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 3 | 2 | 5 | 4 | 6 | NA | NA | NA | NA | NA
Amylase increased (Investigations) | 0 | 0 | 1 | 4 | 1 | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 3 | 7 | 10 | NA | NA | NA | NA | NA
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 3 | 1 | NA | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1 | 3 | 4 | NA | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 2 | 2 | 2 | 8 | 4 | NA | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 3 | 2 | 3 | 5 | 0 | NA | NA | NA | NA | NA
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Lipase increased (Investigations) | 0 | 0 | 2 | 6 | 1 | NA | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | NA | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 1 | 1 | 1 | 2 | 1 | NA | NA | NA | NA | NA
Weight decreased (Investigations) | 2 | 0 | 1 | 2 | 1 | NA | NA | NA | NA | NA
Weight increased (Investigations) | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 3 | 15 | 3 | NA | NA | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 3 | 9 | 4 | NA | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4 | 1 | NA | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 2 | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 5 | 3 | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 3 | 3 | NA | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | NA | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3 | 1 | NA | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 3 | 0 | NA | NA | NA | NA | NA
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 0 | 0 | 0 | 5 | 3 | NA | NA | NA | NA | NA
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Serotonin syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Depression (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 3 | 4 | NA | NA | NA | NA | NA
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 5 | 2 | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 4 | 1 | NA | NA | NA | NA | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | NA | NA | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 4 | 4 | 8 | NA | NA | NA | NA | NA
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 4 | 4 | NA | NA | NA | NA | NA
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 0 | NA | NA | NA | NA | NA
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | NA | NA | NA | NA | NA
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA
Haematoma (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 2 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT02795429/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT02795429/SAP_001.pdf